CLINICAL TRIAL: NCT00732277
Title: Evaluation of Corticosteroid Therapy in Childhood Severe Sepsis (Steroids in Paediatric Sepsis, StePS) - a Randomised Pilot Study
Brief Title: Evaluation of Corticosteroid Therapy in Childhood Severe Sepsis - a Randomised Pilot Study
Acronym: StePS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); St Mary's NHS Trust (Other Government); University of Bristol (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHM CHI 434; 2007-002788-28 (EudraCT Number); 07/H0504/139 (Other: Southampton & South West Hampshire REC)
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Sepsis
Keywords: sepsis; septicaemia; septicemia; paediatric; pediatric; children
MeSH Terms: conditions — Sepsis; Toxemia | interventions — Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Patients in this arm will be given the following IMP intraveneously at 6 hour intervals - hydrocortisone (100mg/m2/24 hours)
  Interventions: Drug: hydrocortisone
- Control (No Intervention): in each phase of study 15 patients will receive no IMP as control arm

INTERVENTIONS:
Drug: hydrocortisone — Patients will be assigned to treatment with hydrocortisone at 100mg/m2/24 hours in 4 divided doses (25 mg/m2/q 6 hourly) for 8 doses (48 hours) in phase 1 of study (45 patients, 30 receive IMP) or 20 doses (120 hours) in phase 2 (45 patients, 30 receive IMP).
  Other Names: Solu-Cortef®; Hydrocortisone sodium succinate
  Arms: Treatment

SUMMARY:
Severe bacterial infections affecting multiple body organs, called severe sepsis (including meningococcal sepsis), remain an important cause of death and disability among children. Although early recognition, powerful antibiotics, and good intensive care have improved outcome, we need new ways to further reduce the number of deaths. Research in adults has shown that steroid replacement therapy might be useful. However, children are known to respond differently to adults and a definitive trial in children is needed because of the potentially harmful as well as beneficial effects of steroids.

This pilot study will provide the necessary information to allow the rational design of a large trial conducted at multiple hospitals investigating the role of corticosteroid replacement therapy in childhood sepsis. The study will provide information on how to measure the effects of steroids, information on length of therapy and a better understanding of how steroids work in children. The results emerging from this study will ultimately allow paediatric intensive care clinicians to know whether or not steroids are safe and/or useful.

The primary objective of this open-label study is therefore to gather clinical and laboratory data with which to inform the design of a large phase 3 double blind randomised controlled trial (RCT). The study will provide basic limited safety data, information on length of therapy and an assessment of possible clinical and laboratory endpoints to be used in addition to mortality.

Definition of sepsis:

Presence of a documented infection (eg clinical evidence of pneumonia, skin or soft tissue infection, purpura fulminans, urinary tract infection, abdominal infection) or a diagnostic positive blood culture (community or hospital acquired) within the last 72 hours and at least two of the following, one of which must be abnormal temperature or leucocyte count[3] core temperature of >38.5°C or <36°C; tachycardia (mean heart rate >2 SD above normal for age); mean respiratory rate > 2 SD above normal for age; leucocyte count elevated or depressed for age.

Definition of severe sepsis:

Sepsis plus cardiovascular organ dysfunction (the need for at least 5mcg/kg/min dopamine or dobutamine, or any amount of adrenaline or noradrenaline support), acute respiratory distress syndrome (ARDS), or 2 or more other organ dysfunctions.

DETAILED DESCRIPTION:
1. PURPOSE: The Need for a Paediatric Trial of Steroids in Sepsis - potential benefits and risks Numerous targets for new therapies in sepsis have been identified, none of which have been shown to have been of benefit in children. The results of adult studies cannot therefore be extrapolated directly to childhood disease. Corticosteroids alter the inflammatory balance in both beneficial and harmful ways in severe sepsis. Recent adult studies have demonstrated transient adrenal insufficiency is associated with adverse outcome and that corticosteroids increase survival in specific patient groups, and steroid replacement has become a standard of care. There is little uniformity in the approach to steroid replacement therapy amongst leading paediatric centres in the UK. Expert opinion has emphasised that guidance is interim while awaiting appropriate paediatric studies. Steroids are perceived as "safe" and "cheap" but should not be introduced into paediatric practice without further research. Sepsis in childhood differs in terms of mortality (around 10% overall in children vs in excess of 40% in adults), background immunity, co-morbidity, and causative organisms. Given the lower overall mortality in childhood sepsis, steroids have the potential to disrupt the inflammatory balance in children causing greater harm than benefit. It is not known which patients should be targeted for therapeutic intervention; what are the most appropriate endpoints; whether the length of steroid therapy can be shorter in children; or whether immunological rebound will occur.
2. DESIGN and METHODOLOGY:

This is an open randomised prospective pilot exploratory study of corticosteroid replacement therapy in three centres. Adrenal function measurements will be assessed on entry to the study. To investigate the inflammatory profile and the impact of corticosteroid replacement, blood will be taken for cytokine and coagulation protein analysis. This study will provide the pilot data necessary for the design of a definitive trial of corticosteroid replacement therapy with the identification of variables likely to improve our ability to stratify patients for intervention and the mechanistic characterisation of the modulatory effects of steroids on inflammation in children with severe sepsis. Enrolment will be undertaken in two stages (see flowsheet diagrams in protocol). Forty five eligible children will be randomly allocated to steroid replacement therapy for 2 days (n=30) or intensive investigation without intervention (n=15) in a 2:1 randomisation (stage 1); 45 subjects (stage 2) will then be randomly allocated to steroid replacement therapy for 5 days (n=30) or intensive investigation without intervention (n=15). Randomisation will the undertaken in accordance with a computer-generated list and will be stratified by age (<1 years; 1 year or more). Progression from stage 1 to stage 2 will follow an interim analysis by a Trial Monitoring Group to ensure safety. This escalating approach will provide safety data, information on length of therapy and an assessment of possible clinical and laboratory endpoints in addition to mortality, reducing the potential for adverse events in the pilot phase while providing data relevant to this population. A large excess of serious adverse events in stage 1 will result in study termination. After careful consideration by the investigators and during the peer review process, placebo will not be used in this study, which will inform a future large phase 3 randomised controlled trial.

RESEARCH PARTICIPANTS WILL RECEIVE THE FOLLOWING INTERVENTIONS THAT ARE NOT PART OF ROUTINE CLINICAL CARE (Please also refer to figures 1-4 in the protocol that we are unable to reproduce here): Children will be screened on admission to PICU. Entry into the study following consent involves a clinical test of endocrine function involving 2 blood tests. The list of procedures conducted in the study is as follows:

1. confirm eligibility requirements, assess pre-existing conditions and medical history, record weight, height, vital signs, data to inform clinical severity scores, complete infection assessment, clinically relevant laboratory investigations
2. corticotrophin stimulation test
3. multiple study samples (endocrine, cytokine and coagulation tests)
4. corticosteroid treatment if randomised to treatment group
5. follow-up in routine clinic

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis where enrolment can occur within 20 hours of first contact with paediatric intensive care, or within 20 hours of the diagnosis of severe sepsis when this diagnosis is made on PICU. Randomisation should occur within 24 hours of first contact with paediatric intensive care, or within 24 hours of the diagnosis of severe sepsis when this diagnosis is made on PICU.
* Requiring mechanical ventilation (The subjects must be mechanically ventilated for entry into the study but this is not time limited. It is routine practice at study centres to pre-emptively ventilate children with evolving sepsis)

Exclusion Criteria:

* Concomitant steroid therapy, vasopressor treatment >24 hrs or use of etomidate (not recommended for use in children less than 10 years and selectively inhibits 11 beta-hydroxylase)
* Patients who have a recognised indication for steroids
* Other immunosuppressive/immunomodulatory therapy (not including intravenous immunoglobulin which is considered standard therapy in toxic shock syndrome and may be given for this indication)
* Significant immunocompromise (eg HIV infection)
* Advanced malignancy
* Burns
* Cardiopulmonary resuscitation
* Children not likely to survive the time period of the maximum study intervention (5 days)
* Patients who have undergone organ transplantation (including bone marrow transplantation)
* Patients undergoing plasma exchange or whole blood exchange transfusion
* Treatment with an investigational drug or device within the last 30 days prior to enrolment.
* Patients who have experienced a prior episode of infection or sepsis during the current hospitalisation.
* Patients who are pregnant (a pregnancy test will be carried out for females of 11 years and above as is standard practice for clinical trials).
* Immediate families of investigators or site personnel directly affiliated with the study. Immediate family is defined as child or sibling, whether biological or legally adopted.

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
primary efficacy endpoint is all cause mortality | 28 days
primary toxicity endpoint is Serious Adverse Events, excluding sepsis-related events specified as secondary outcomes | 28 days

SECONDARY OUTCOMES:
PIM2 | entry
PELOD | daily to 28 days or PICU discharge
ICU mortality | 28 days
time until shock reversal, defined as cessation of inotropic support for 24 hours | 28 days
time to resolution of multiorgan dysfunction | 28 days
time to resolution of base deficit | 28 days
time to resolution of lactate | 28 days
time to decision to discharge from ICU | 28 days
laboratory analysis of adrenal function | 6 days and convalescence
laboratory analysis of inflammatory parameters (defined in protocol) | 6 days and convalescence
laboratory analysis of coagulation parameters (defined in protocol) | 6 days and convalescence

CONTACTS AND LOCATIONS:
Overall Officials: Saul N Faust, MBBS PhD, Study Chair — University of Southampton; Simon Nadel, MB BS, Principal Investigator — Imperial College London; Robert S Heyderman, MBBS PhD, Study Director — University of Liverpool; Diana M Gibb, MBChB MD, Study Director — Medical Research Council; Michael Levin, MBBCH PhD, Study Director — Imperial College London; Andrew Wolf, MBBChir MD, Principal Investigator — Univeristy of Bristol; John V Pappachan, MB BChir, Study Director — University Hospital Southampton NHS Foundation Trust; Sarah Walker, MA PhD, Study Director — Medical Research Council; Carrol Gamble, PhD, Study Director — University of Liverpool / MCRN Clinical Trials Unit
Locations (3):
- United Kingdom (3):
  - Bristol Royal Hospital for Children, Bristol, UK
  - Imperial College Healthcare NHS Trust, London, UK
  - Southampton University Hospitals NHS Trust, Southampton, UK

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aneja R, Carcillo JA. What is the rationale for hydrocortisone treatment in children with infection-related adrenal insufficiency and septic shock? Arch Dis Child. 2007 Feb;92(2):165-9. doi: 10.1136/adc.2005.088450. Epub 2006 Sep 26. PMID 17003064
- [Background] Booy R, Habibi P, Nadel S, de Munter C, Britto J, Morrison A, Levin M; Meningococcal Research Group. Reduction in case fatality rate from meningococcal disease associated with improved healthcare delivery. Arch Dis Child. 2001 Nov;85(5):386-90. doi: 10.1136/adc.85.5.386. PMID 11668100
- [Background] Despond O, Proulx F, Carcillo JA, Lacroix J. Pediatric sepsis and multiple organ dysfunction syndrome. Curr Opin Pediatr. 2001 Jun;13(3):247-53. doi: 10.1097/00008480-200106000-00006. PMID 11389359
- [Background] Stoll BJ, Holman RC, Schuchat A. Decline in sepsis-associated neonatal and infant deaths in the United States, 1979 through 1994. Pediatrics. 1998 Aug;102(2):e18. doi: 10.1542/peds.102.2.e18. PMID 9685463
- [Background] Thorburn K, Baines P, Thomson A, Hart CA. Mortality in severe meningococcal disease. Arch Dis Child. 2001 Nov;85(5):382-5. doi: 10.1136/adc.85.5.382. PMID 11668098
- [Background] Watson RS, Carcillo JA, Linde-Zwirble WT, Clermont G, Lidicker J, Angus DC. The epidemiology of severe sepsis in children in the United States. Am J Respir Crit Care Med. 2003 Mar 1;167(5):695-701. doi: 10.1164/rccm.200207-682OC. Epub 2002 Nov 14. PMID 12433670
- [Background] Cohen J. The immunopathogenesis of sepsis. Nature. 2002 Dec 19-26;420(6917):885-91. doi: 10.1038/nature01326. PMID 12490963
- [Background] Boldrick JC, Alizadeh AA, Diehn M, Dudoit S, Liu CL, Belcher CE, Botstein D, Staudt LM, Brown PO, Relman DA. Stereotyped and specific gene expression programs in human innate immune responses to bacteria. Proc Natl Acad Sci U S A. 2002 Jan 22;99(2):972-7. doi: 10.1073/pnas.231625398. PMID 11805339
- [Background] Nau GJ, Richmond JF, Schlesinger A, Jennings EG, Lander ES, Young RA. Human macrophage activation programs induced by bacterial pathogens. Proc Natl Acad Sci U S A. 2002 Feb 5;99(3):1503-8. doi: 10.1073/pnas.022649799. Epub 2002 Jan 22. PMID 11805289
- [Background] Faust SN, Heyderman RS, Levin M. Disseminated intravascular coagulation and purpura fulminans secondary to infection. Baillieres Best Pract Res Clin Haematol. 2000 Jun;13(2):179-97. doi: 10.1053/beha.2000.0067. PMID 10942620
- [Background] Bone RC, Grodzin CJ, Balk RA. Sepsis: a new hypothesis for pathogenesis of the disease process. Chest. 1997 Jul;112(1):235-43. doi: 10.1378/chest.112.1.235. No abstract available. PMID 9228382
- [Background] van Dissel JT, van Langevelde P, Westendorp RG, Kwappenberg K, Frolich M. Anti-inflammatory cytokine profile and mortality in febrile patients. Lancet. 1998 Mar 28;351(9107):950-3. doi: 10.1016/S0140-6736(05)60606-X. PMID 9734942
- [Background] Hotchkiss RS, Swanson PE, Freeman BD, Tinsley KW, Cobb JP, Matuschak GM, Buchman TG, Karl IE. Apoptotic cell death in patients with sepsis, shock, and multiple organ dysfunction. Crit Care Med. 1999 Jul;27(7):1230-51. doi: 10.1097/00003246-199907000-00002. PMID 10446814
- [Background] Hibberd ML, Sumiya M, Summerfield JA, Booy R, Levin M. Association of variants of the gene for mannose-binding lectin with susceptibility to meningococcal disease. Meningococcal Research Group. Lancet. 1999 Mar 27;353(9158):1049-53. doi: 10.1016/s0140-6736(98)08350-0. PMID 10199352
- [Background] Nadel S, Newport MJ, Booy R, Levin M. Variation in the tumor necrosis factor-alpha gene promoter region may be associated with death from meningococcal disease. J Infect Dis. 1996 Oct;174(4):878-80. doi: 10.1093/infdis/174.4.878. PMID 8843235
- [Background] Arnalich F, Lopez-Maderuelo D, Codoceo R, Lopez J, Solis-Garrido LM, Capiscol C, Fernandez-Capitan C, Madero R, Montiel C. Interleukin-1 receptor antagonist gene polymorphism and mortality in patients with severe sepsis. Clin Exp Immunol. 2002 Feb;127(2):331-6. doi: 10.1046/j.1365-2249.2002.01743.x. PMID 11876758
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Bernard GR, Vincent JL, Laterre PF, LaRosa SP, Dhainaut JF, Lopez-Rodriguez A, Steingrub JS, Garber GE, Helterbrand JD, Ely EW, Fisher CJ Jr; Recombinant human protein C Worldwide Evaluation in Severe Sepsis (PROWESS) study group. Efficacy and safety of recombinant human activated protein C for severe sepsis. N Engl J Med. 2001 Mar 8;344(10):699-709. doi: 10.1056/NEJM200103083441001. PMID 11236773
- [Background] Marik PE, Zaloga GP. Adrenal insufficiency in the critically ill: a new look at an old problem. Chest. 2002 Nov;122(5):1784-96. doi: 10.1378/chest.122.5.1784. PMID 12426284
- [Background] Bone RC, Fisher CJ Jr, Clemmer TP, Slotman GJ, Metz CA, Balk RA. A controlled clinical trial of high-dose methylprednisolone in the treatment of severe sepsis and septic shock. N Engl J Med. 1987 Sep 10;317(11):653-8. doi: 10.1056/NEJM198709103171101. PMID 3306374
- [Background] Sprung CL, Caralis PV, Marcial EH, Pierce M, Gelbard MA, Long WM, Duncan RC, Tendler MD, Karpf M. The effects of high-dose corticosteroids in patients with septic shock. A prospective, controlled study. N Engl J Med. 1984 Nov 1;311(18):1137-43. doi: 10.1056/NEJM198411013111801. PMID 6384785
- [Background] Cronin L, Cook DJ, Carlet J, Heyland DK, King D, Lansang MA, Fisher CJ Jr. Corticosteroid treatment for sepsis: a critical appraisal and meta-analysis of the literature. Crit Care Med. 1995 Aug;23(8):1430-9. doi: 10.1097/00003246-199508000-00019. PMID 7634816
- [Background] Bollaert PE, Fieux F, Charpentier C, Levy B. Baseline cortisol levels, cortisol response to corticotropin, and prognosis in late septic shock. Shock. 2003 Jan;19(1):13-5. doi: 10.1097/00024382-200301000-00003. PMID 12558137
- [Background] Hatherill M, Tibby SM, Hilliard T, Turner C, Murdoch IA. Adrenal insufficiency in septic shock. Arch Dis Child. 1999 Jan;80(1):51-5. doi: 10.1136/adc.80.1.51. PMID 10325759
- [Background] van Woensel JB, Biezeveld MH, Alders AM, Eerenberg AJ, Endert E, Hack EC, von Rosenstiel IA, Kuijpers TW. Adrenocorticotropic hormone and cortisol levels in relation to inflammatory response and disease severity in children with meningococcal disease. J Infect Dis. 2001 Dec 15;184(12):1532-7. doi: 10.1086/324673. Epub 2001 Dec 3. PMID 11740728
- [Background] Marik PE, Zaloga GP. Adrenal insufficiency during septic shock. Crit Care Med. 2003 Jan;31(1):141-5. doi: 10.1097/00003246-200301000-00022. PMID 12545007
- [Background] Annane D, Sebille V, Troche G, Raphael JC, Gajdos P, Bellissant E. A 3-level prognostic classification in septic shock based on cortisol levels and cortisol response to corticotropin. JAMA. 2000 Feb 23;283(8):1038-45. doi: 10.1001/jama.283.8.1038. PMID 10697064
- [Background] Pizarro CF, Troster EJ, Damiani D, Carcillo JA. Absolute and relative adrenal insufficiency in children with septic shock. Crit Care Med. 2005 Apr;33(4):855-9. doi: 10.1097/01.ccm.0000159854.23324.84. PMID 15818116
- [Background] Bollaert PE, Charpentier C, Levy B, Debouverie M, Audibert G, Larcan A. Reversal of late septic shock with supraphysiologic doses of hydrocortisone. Crit Care Med. 1998 Apr;26(4):645-50. doi: 10.1097/00003246-199804000-00010. PMID 9559600
- [Background] Briegel J, Forst H, Haller M, Schelling G, Kilger E, Kuprat G, Hemmer B, Hummel T, Lenhart A, Heyduck M, Stoll C, Peter K. Stress doses of hydrocortisone reverse hyperdynamic septic shock: a prospective, randomized, double-blind, single-center study. Crit Care Med. 1999 Apr;27(4):723-32. doi: 10.1097/00003246-199904000-00025. PMID 10321661
- [Background] Briegel J, Kellermann W, Forst H, Haller M, Bittl M, Hoffmann GE, Buchler M, Uhl W, Peter K. Low-dose hydrocortisone infusion attenuates the systemic inflammatory response syndrome. The Phospholipase A2 Study Group. Clin Investig. 1994 Oct;72(10):782-7. doi: 10.1007/BF00180547. PMID 7865982
- [Background] Keh D, Boehnke T, Weber-Cartens S, Schulz C, Ahlers O, Bercker S, Volk HD, Doecke WD, Falke KJ, Gerlach H. Immunologic and hemodynamic effects of "low-dose" hydrocortisone in septic shock: a double-blind, randomized, placebo-controlled, crossover study. Am J Respir Crit Care Med. 2003 Feb 15;167(4):512-20. doi: 10.1164/rccm.200205-446OC. Epub 2002 Nov 8. PMID 12426230
- [Background] Leone M, Boutiere-Albanese B, Valette S, Camoin-Jau L, Barrau K, Albanese J, Martin C, Dignat-George F. Cell adhesion molecules as a marker reflecting the reduction of endothelial activation induced by glucocorticoids. Shock. 2004 Apr;21(4):311-4. doi: 10.1097/00024382-200404000-00004. PMID 15179130
- [Background] Maxime V, Fitting C, Annane D, Cavaillon JM. Corticoids normalize leukocyte production of macrophage migration inhibitory factor in septic shock. J Infect Dis. 2005 Jan 1;191(1):138-44. doi: 10.1086/426401. Epub 2004 Nov 30. PMID 15593015
- [Background] Mussack T, Briegel J, Schelling G, Biberthaler P, Jochum M. Effect of stress doses of hydrocortisone on S-100B vs. interleukin-8 and polymorphonuclear elastase levels in human septic shock. Clin Chem Lab Med. 2005;43(3):259-68. doi: 10.1515/CCLM.2005.044. PMID 15843228
- [Background] Oppert M, Schindler R, Husung C, Offermann K, Graf KJ, Boenisch O, Barckow D, Frei U, Eckardt KU. Low-dose hydrocortisone improves shock reversal and reduces cytokine levels in early hyperdynamic septic shock. Crit Care Med. 2005 Nov;33(11):2457-64. doi: 10.1097/01.ccm.0000186370.78639.23. PMID 16276166
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Background] Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for severe sepsis and septic shock: a systematic review and meta-analysis. BMJ. 2004 Aug 28;329(7464):480. doi: 10.1136/bmj.38181.482222.55. Epub 2004 Aug 2. PMID 15289273
- [Background] Minneci PC, Deans KJ, Banks SM, Eichacker PQ, Natanson C. Meta-analysis: the effect of steroids on survival and shock during sepsis depends on the dose. Ann Intern Med. 2004 Jul 6;141(1):47-56. doi: 10.7326/0003-4819-141-1-200407060-00014. PMID 15238370
- [Background] Prigent H, Maxime V, Annane D. Clinical review: corticotherapy in sepsis. Crit Care. 2004 Apr;8(2):122-9. doi: 10.1186/cc2374. Epub 2003 Sep 29. PMID 15025773
- [Background] Keh D, Sprung CL. Use of corticosteroid therapy in patients with sepsis and septic shock: an evidence-based review. Crit Care Med. 2004 Nov;32(11 Suppl):S527-33. doi: 10.1097/01.ccm.0000142983.15421.11. PMID 15542960
- [Background] Sessler CN. Steroids for septic shock: back from the dead? (Con). Chest. 2003 May;123(5 Suppl):482S-9S. doi: 10.1378/chest.123.5_suppl.482s. PMID 12740233
- [Background] Fessler MB, O'Brien JM, Douglas IS. Laboratory predictors of relative adrenal insufficiency in septic shock. Crit Care Med. 2003 Aug;31(8):2251-2; author reply 2252-3. doi: 10.1097/01.CCM.0000080486.95472.A3. No abstract available. PMID 12973195
- [Background] Sprung CL, Annane D, Keh D, Moreno R, Singer M, Freivogel K, Weiss YG, Benbenishty J, Kalenka A, Forst H, Laterre PF, Reinhart K, Cuthbertson BH, Payen D, Briegel J; CORTICUS Study Group. Hydrocortisone therapy for patients with septic shock. N Engl J Med. 2008 Jan 10;358(2):111-24. doi: 10.1056/NEJMoa071366. PMID 18184957
- [Background] Nadel S, Goldstein B, Williams MD, Dalton H, Peters M, Macias WL, Abd-Allah SA, Levy H, Angle R, Wang D, Sundin DP, Giroir B; REsearching severe Sepsis and Organ dysfunction in children: a gLobal perspective (RESOLVE) study group. Drotrecogin alfa (activated) in children with severe sepsis: a multicentre phase III randomised controlled trial. Lancet. 2007 Mar 10;369(9564):836-843. doi: 10.1016/S0140-6736(07)60411-5. PMID 17350452
- [Background] Hildebrandt T, Mansour M, Al Samsam R. The use of steroids in children with septicemia: review of the literature and assessment of current practice in PICUs in the UK. Paediatr Anaesth. 2005 May;15(5):358-65. doi: 10.1111/j.1460-9592.2004.01540.x. No abstract available. PMID 15828985
- [Background] Branco RG, Russell RR. Should steroids be used in children with meningococcal shock? Arch Dis Child. 2005 Nov;90(11):1195-6. doi: 10.1136/adc.2005.077701. No abstract available. PMID 16243881
- [Background] Carcillo JA, Fields AI; American College of Critical Care Medicine Task Force Committee Members. Clinical practice parameters for hemodynamic support of pediatric and neonatal patients in septic shock. Crit Care Med. 2002 Jun;30(6):1365-78. doi: 10.1097/00003246-200206000-00040. PMID 12072696
- [Background] Kleinman ME. Clinical practice parameters for pediatric and neonatal septic shock: to have or to have not? Crit Care Med. 2002 Jun;30(6):1400-1. doi: 10.1097/00003246-200206000-00056. No abstract available. PMID 12072711
- [Background] Parker MM, Hazelzet JA, Carcillo JA. Pediatric considerations. Crit Care Med. 2004 Nov;32(11 Suppl):S591-4. doi: 10.1097/01.ccm.0000145904.97821.0d. PMID 15542968
- [Background] Feezor RJ, Cheng A, Paddock HN, Baker HV, Moldawer LL. Functional genomics and gene expression profiling in sepsis: beyond class prediction. Clin Infect Dis. 2005 Nov 15;41 Suppl 7:S427-35. doi: 10.1086/431993. PMID 16237642
- [Background] Proulx F, Fayon M, Farrell CA, Lacroix J, Gauthier M. Epidemiology of sepsis and multiple organ dysfunction syndrome in children. Chest. 1996 Apr;109(4):1033-7. doi: 10.1378/chest.109.4.1033. PMID 8635327
- [Background] Barsness KA, Bensard DD, Partrick DA, Calkins CM, Hendrickson RJ, McIntyre RC Jr. Endotoxin induces an exaggerated interleukin-10 response in peritoneal macrophages of children compared with adults. J Pediatr Surg. 2004 Jun;39(6):912-5; discussion 912-5. doi: 10.1016/j.jpedsurg.2004.02.009. PMID 15185224
- [Background] Johnston JA, Yi MS, Britto MT, Mrus JM. Importance of organ dysfunction in determining hospital outcomes in children. J Pediatr. 2004 May;144(5):595-601. doi: 10.1016/j.jpeds.2004.01.045. PMID 15126992
- [Background] Slater A, Shann F, Pearson G; Paediatric Index of Mortality (PIM) Study Group. PIM2: a revised version of the Paediatric Index of Mortality. Intensive Care Med. 2003 Feb;29(2):278-85. doi: 10.1007/s00134-002-1601-2. Epub 2003 Jan 23. PMID 12541154
- [Background] Leteurtre S, Duhamel A, Grandbastien B, Lacroix J, Leclerc F. Paediatric logistic organ dysfunction (PELOD) score. Lancet. 2006 Mar 18;367(9514):897; author reply 900-2. doi: 10.1016/S0140-6736(06)68371-2. No abstract available. PMID 16546531
- [Background] Leteurtre S, Martinot A, Duhamel A, Proulx F, Grandbastien B, Cotting J, Gottesman R, Joffe A, Pfenninger J, Hubert P, Lacroix J, Leclerc F. Validation of the paediatric logistic organ dysfunction (PELOD) score: prospective, observational, multicentre study. Lancet. 2003 Jul 19;362(9379):192-7. doi: 10.1016/S0140-6736(03)13908-6. PMID 12885479
- [Background] Vogeser M, Groetzner J, Kupper C, Briegel J. Free serum cortisol during the postoperative acute phase response determined by equilibrium dialysis liquid chromatography-tandem mass spectrometry. Clin Chem Lab Med. 2003 Feb;41(2):146-51. doi: 10.1515/CCLM.2003.024. PMID 12666999
- [Background] Hamrahian AH, Oseni TS, Arafah BM. Measurements of serum free cortisol in critically ill patients. N Engl J Med. 2004 Apr 15;350(16):1629-38. doi: 10.1056/NEJMoa020266. PMID 15084695
- [Background] Arlt W, Hammer F, Sanning P, Butcher SK, Lord JM, Allolio B, Annane D, Stewart PM. Dissociation of serum dehydroepiandrosterone and dehydroepiandrosterone sulfate in septic shock. J Clin Endocrinol Metab. 2006 Jul;91(7):2548-54. doi: 10.1210/jc.2005-2258. Epub 2006 Apr 11. PMID 16608898
- [Background] Yu SL, Chen HW, Yang PC, Peck K, Tsai MH, Chen JJ, Lin FY. Differential gene expression in gram-negative and gram-positive sepsis. Am J Respir Crit Care Med. 2004 May 15;169(10):1135-43. doi: 10.1164/rccm.200211-1278OC. Epub 2004 Mar 4. PMID 15001460
- [Background] Dorn LD, Lucke JF, Loucks TL, Berga SL. Salivary cortisol reflects serum cortisol: analysis of circadian profiles. Ann Clin Biochem. 2007 May;44(Pt 3):281-4. doi: 10.1258/000456307780480954. PMID 17456296
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637
- [Background] Wetherell MA, Crown AL, Lightman SL, Miles JN, Kaye J, Vedhara K. The four-dimensional stress test: psychological, sympathetic-adrenal-medullary, parasympathetic and hypothalamic-pituitary-adrenal responses following inhalation of 35% CO2. Psychoneuroendocrinology. 2006 Jul;31(6):736-47. doi: 10.1016/j.psyneuen.2006.02.005. Epub 2006 Apr 18. PMID 16621326
- [Background] Faust SN, Levin M, Harrison OB, Goldin RD, Lockhart MS, Kondaveeti S, Laszik Z, Esmon CT, Heyderman RS. Dysfunction of endothelial protein C activation in severe meningococcal sepsis. N Engl J Med. 2001 Aug 9;345(6):408-16. doi: 10.1056/NEJM200108093450603. PMID 11496851
- [Background] Pathan N, Hemingway CA, Alizadeh AA, Stephens AC, Boldrick JC, Oragui EE, McCabe C, Welch SB, Whitney A, O'Gara P, Nadel S, Relman DA, Harding SE, Levin M. Role of interleukin 6 in myocardial dysfunction of meningococcal septic shock. Lancet. 2004 Jan 17;363(9404):203-9. doi: 10.1016/S0140-6736(03)15326-3. PMID 14738793
- [Background] Heyderman RS, Ison CA, Peakman M, Levin M, Klein NJ. Neutrophil response to Neisseria meningitidis: inhibition of adhesion molecule expression and phagocytosis by recombinant bactericidal/permeability-increasing protein (rBPI21). J Infect Dis. 1999 May;179(5):1288-92. doi: 10.1086/314706. PMID 10191239
- [Background] Klein NJ, Ison CA, Peakman M, Levin M, Hammerschmidt S, Frosch M, Heyderman RS. The influence of capsulation and lipooligosaccharide structure on neutrophil adhesion molecule expression and endothelial injury by Neisseria meningitidis. J Infect Dis. 1996 Jan;173(1):172-9. doi: 10.1093/infdis/173.1.172. PMID 8537655
- [Background] Ison CA, Heyderman RS, Klein NJ, Peakman M, Levin M. Whole blood model of meningococcal bacteraemia--a method for exploring host-bacterial interactions. Microb Pathog. 1995 Feb;18(2):97-107. doi: 10.1016/s0882-4010(95)90093-4. PMID 7643746
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Background] Luscombe M, Owens B. Weight estimation in resuscitation: is the current formula still valid? Arch Dis Child. 2007 May;92(5):412-5. doi: 10.1136/adc.2006.107284. Epub 2007 Jan 9. PMID 17213259
- [Background] Bellomo R, McGrath B, Boyce N. Effect of continuous venovenous hemofiltration with dialysis on hormone and catecholamine clearance in critically ill patients with acute renal failure. Crit Care Med. 1994 May;22(5):833-7. doi: 10.1097/00003246-199405000-00020. PMID 8181293
- [Background] Derkx B, Wittes J, McCloskey R. Randomized, placebo-controlled trial of HA-1A, a human monoclonal antibody to endotoxin, in children with meningococcal septic shock. European Pediatric Meningococcal Septic Shock Trial Study Group. Clin Infect Dis. 1999 Apr;28(4):770-7. doi: 10.1086/515184. PMID 10825037
- [Background] Levin M, Quint PA, Goldstein B, Barton P, Bradley JS, Shemie SD, Yeh T, Kim SS, Cafaro DP, Scannon PJ, Giroir BP. Recombinant bactericidal/permeability-increasing protein (rBPI21) as adjunctive treatment for children with severe meningococcal sepsis: a randomised trial. rBPI21 Meningococcal Sepsis Study Group. Lancet. 2000 Sep 16;356(9234):961-7. doi: 10.1016/s0140-6736(00)02712-4. PMID 11041396
- [Background] Barton P, Kalil AC, Nadel S, Goldstein B, Okhuysen-Cawley R, Brilli RJ, Takano JS, Martin LD, Quint P, Yeh TS, Dalton HJ, Gessouron MR, Brown KE, Betts H, Levin M, Macias WL, Small DS, Wyss VL, Bates BM, Utterback BG, Giroir BP. Safety, pharmacokinetics, and pharmacodynamics of drotrecogin alfa (activated) in children with severe sepsis. Pediatrics. 2004 Jan;113(1 Pt 1):7-17. doi: 10.1542/peds.113.1.7. PMID 14702440
- [Background] Humphreys N, Bays SM, Parry AJ, Pawade A, Heyderman RS, Wolf AR. Spinal anesthesia with an indwelling catheter reduces the stress response in pediatric open heart surgery. Anesthesiology. 2005 Dec;103(6):1113-20. doi: 10.1097/00000542-200512000-00003. PMID 16306721
- [Background] Weale NK, Rogers CA, Cooper R, Nolan J, Wolf AR. Effect of remifentanil infusion rate on stress response to the pre-bypass phase of paediatric cardiac surgery. Br J Anaesth. 2004 Feb;92(2):187-94. doi: 10.1093/bja/aeh038. PMID 14722167
- [Background] Duncan HP, Cloote A, Weir PM, Jenkins I, Murphy PJ, Pawade AK, Rogers CA, Wolf AR. Reducing stress responses in the pre-bypass phase of open heart surgery in infants and young children: a comparison of different fentanyl doses. Br J Anaesth. 2000 May;84(5):556-64. doi: 10.1093/bja/84.5.556. PMID 10844829
- See also: UK NIHR Medicines For Children Research Network — http://www.mcrn.org.uk/